CLINICAL TRIAL: NCT02168686
Title: Phase 1/2 Study of Intravenous or Intrapleural Administration of a Serotype rh.10 Replication Deficient Adeno-associated Virus Gene Transfer Vector Expressing the Human Alpha-1 Antitrypsin cDNA to Individuals With Alpha-1 Antitrypsin Deficiency
Brief Title: Safety Dose Finding Study of ADVM-043 Gene Therapy to Treat Alpha-1 Antitrypsin (A1AT) Deficiency
Acronym: ADVANCE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Adverum Biotechnologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADVM-043-01
Record Dates: First submitted 2014-06-10; First posted 2014-06-20 (Estimated); Results first posted 2022-08-08 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Alpha 1-Antitrypsin Deficiency
Keywords: alpha-1 antitrypsin deficiency; alpha1-antitrypsin deficiency; alpha-1-antitrypsin deficiency; alpha1AT; A1AT; ADVM-043; AAVrh.10halpha1AT; AAVrh.10hA1AT; Gene transfer vector; Gene therapy; Lung disease; Emphysema; COPD; ADVANCE study; ADVM-043-01
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Lung Diseases; Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Open-label, multicenter, dose-escalation clinical study to assess the safety and treatment effect of ADVM-043 in subjects with Alpha-1 Antitrypsin Deficiency.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A: Dose 1 (Experimental): ADVM-043, at the lowest dose of three planned dose levels, of 8E13 total vg (equivalent to 1E12 vg/kg based on an 80-kg patient) administered IV
  Interventions: Genetic: ADVM-043
- Part A: Dose 2 (Experimental): ADVM-043 at the intermediate dose of three planned dose levels, of 4E14 total vg (equivalent to 5E12 vg/kg based on an 80-kg patient) administered IV
  Interventions: Genetic: ADVM-043
- Part A: Dose 3 (Experimental): ADVM-043 at the highest dose of three planned dose levels, of 1.2E15 total vg (equivalent to 1.5E13 vg/kg based on an 80-kg patient) administered IV
  Interventions: Genetic: ADVM-043
- Part A: Dose 4 (Experimental): ADVM-043 administered at a dose that will be determined
  Interventions: Genetic: ADVM-043
- Part B (optional): Intrapleural administration (Experimental): ADVM-043 administered intrapleurally at a dose that will be determined
  Interventions: Genetic: ADVM-043

INTERVENTIONS:
Genetic: ADVM-043 — Gene transfer vector administration
  Other Names: AAVrh.10halpha1AT; AAVrh.10hA1AT

SUMMARY:
The ADVANCE study is being conducted by Adverum Biotechnologies, Inc. as an open-label, multicenter, dose-escalation study in order to assess the safety and protein expression of ADVM-043 following a single intravenous or intrapleural administration.

DETAILED DESCRIPTION:
Alpha-1 Antitrypsin (A1AT) is a major inhibitor of serine proteases and plays an important role in the lung as an inhibitor of neutrophil elastase. A1AT deficiency is associated with decreases in plasma A1AT levels and is associated with an increased risk for developing asthma, emphysema/COPD, and bronchiectasis. Much of the lung damage is thought to be caused by proteolytic damage from neutrophil elastase and other proteases.

ADVM-043 is an investigational gene therapy product (serotype AAVrh.10 vector) expressing human A1AT that is intended to deliver a functional gene to the liver of patients with A1AT deficiency. Study ADVM-043-01 will study up to 4 dose levels in up to 20 patients and assess the hypothesis that a single administration of an AAV vector expressing the human M-type A1AT (i.e., ADVM-043) to patients with A1AT deficiency is safe and results in persistent therapeutic levels of A1AT in blood and alveolar epithelial lining fluid (epithelial lining fluid is only to be collected in subjects who are dosed intrapleurally). The primary endpoint is safety, and changes in plasma A1AT levels at multiple time points up to 52 weeks after dosing. A prophylactic tapering corticosteroid regimen will be used to protect against potential vector induced transaminitis. Subjects will be followed for up to 52 weeks after dosing. Safety and efficacy data from the IV cohorts will be considered when determining whether to proceed to intrapleural administration. After completion of this study, subjects will be asked to enroll in a Long Term Follow Up study.

ELIGIBILITY:
Key Inclusion Criteria:

* Capable of providing informed consent
* Alpha1AT genotype of ZZ or Z Null
* Males and females 18 years and older
* Ongoing treatment with A1AT augmentation is not required, however any subject receiving A1AT augmentation therapy must be willing to washout. Washout is defined as at least 8 weeks between last augmentation therapy and pre-treatment plasma A1AT level
* Willing to remain off PAT for at least 3 months following treatment
* Body mass index 18 to 35 kg/m2
* Fertile men and women of childbearing potential must agree to use barrier contraception for 3 months after treatment

Key Exclusion Criteria:

* FEV1 <35 percent of predicted value at the Screening visit
* Receiving systemic corticosteroids or other immunosuppressive medications
* Immunodeficiency disease or evidence of active infection of any type, including human immunodeficiency virus
* Abnormal liver function tests
* Organ transplant recipient or awaiting transplantation
* Participation in another current or previous gene transfer study
* AAVrh.10 neutralizing antibody titer ≥ 1:5
* Female who is pregnant or lactating
* History of alcohol or drug abuse within the past 5 years
* Any history of allergies that may prohibit study-specific investigations
* Receiving an investigational medicinal product or participating in another investigational study within 3 months prior to consent
* Cigarette smoking, or any other tobacco use, e-cigarettes or other recreational inhalant within 1 year of the Screening Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charlton Strange, MD, Principal Investigator — Medical University of South Carolina, Charleston, SC, USA; Friedrich Kueppers, MD, Principal Investigator — Temple University Hospital, Philadelphia, PA, USA; Mark Brantly, MD, Principal Investigator — University of Florida, Gainesville, FL, USA; Kyle Hogarth, MD, Principal Investigator — University of Chicago Medical Center, Chicago, IL, USA; Igor Barjakatarevic, MD, Principal Investigator — Ronald Reagan UCLA Medical Center, Santa Monica, CA, USA
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- [Derived] Remih K, Amzou S, Strnad P. Alpha1-antitrypsin deficiency: New therapies on the horizon. Curr Opin Pharmacol. 2021 Aug;59:149-156. doi: 10.1016/j.coph.2021.06.001. Epub 2021 Jul 10. PMID 34256305

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Dose 1: Single IV infusion of ADVM-043 at 8E13 total vg
- Part A: Dose 2: Single IV infusion of ADVM-043 at 4E14 total vg
- Part A: Dose 3: Single IV infusion of ADVM-043 at 1.2E15 total vg
Period: Overall Study
Arm/Group | Part A: Dose 1 | Part A: Dose 2 | Part A: Dose 3
Started | 2 | 2 | 2
Completed | 2 | 2 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Dose 1 | Part A: Dose 2 | Part A: Dose 3 | Total
Number analyzed (Participants) | 2 | 2 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 1 | 5
  >=65 years | 0 | 0 | 1 | 1
Age, Continuous [Mean (Full Range); unit: years] | 40.5 [25 to 56] | 53.5 [52 to 55] | 61.0 [53 to 69] | 51.7 [25 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 3
  Male | 2 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 2 | 2 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Events Related to ADVM-043
Description: Number and proportion of subjects experiencing treatment-related adverse events related to ADVM-043
Time Frame: From ADVM-043 infusion through End-of-Study visit at 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Dose 1 | Part A: Dose 2 | Part A: Dose 3
Number analyzed (Participants) | 2 | 2 | 2
Participants | 0 | 1 | 2

2. Primary Outcome: Abnormal Changes in Clinical Laboratory Parameters
Description: Number of participants with ≥1 abnormal shift from Baseline in neutrophil count, hemoglobin, important serum chemistry parameters
Time Frame: From ADVM-043 infusion through End-of-Study visit at 52 weeks
Measure: Number; unit: participants
Groups:
- Total: All Participants
Arm/Group | Part A: Dose 1 | Part A: Dose 2 | Part A: Dose 3 | Total
Number analyzed (Participants) | 2 | 2 | 2 | 6
participants
  Neutrophil Count Shifts to High | 2 | 1 | 2 | 5
  Neutrophil Count Shifts to Low | 0 | 0 | 0 | 0
  Hemoglobin Shifts to High | 0 | 1 | 1 | 2
  Hemoglobin Shifts to Low | 0 | 0 | 0 | 0
  Alanine Transaminase Shifts to High (max >1.0 to ≤2.0×upper limit of normal) | 1 | 1 | 1 | 3
  Alanine Transaminase Shifts to High (max >2.0 to ≤3.0×upper limit of normal | 0 | 1 | 1 | 2
  Alanine Transaminase Shifts to High (max >3.0×upper limit of normal) | 0 | 0 | 0 | 0
  Aspartate Transaminase Shifts to High (max >1.0 to ≤2.0×upper limit of normal) | 0 | 1 | 1 | 2
  Aspartate Transaminase Shifts to High (max >2.0 to ≤3.0×upper limit of normal) | 0 | 0 | 1 | 1
  Aspartate Transaminase Shifts to High (max >3.0×upper limit of normal) | 0 | 0 | 0 | 0
  Alkaline Phosphatase Shifts to High | 0 | 0 | 1 | 1
  Creatinine Shifts to High | 0 | 0 | 0 | 0
  Creatinine Shifts to Low | 0 | 0 | 1 | 1
  Creatine Kinase Shifts to High | 1 | 0 | 1 | 2
  Creatine Kinase Shifts to Low | 1 | 0 | 0 | 1
  Albumin Shifts to High | 0 | 0 | 0 | 0
  Albumin Shifts to Low | 0 | 0 | 0 | 0
  Direct Bilirubin Shifts to High | 0 | 0 | 0 | 0
  Direct Bilirubin Shifts to Low | 0 | 0 | 0 | 0
  Serum Glucose Shifts to High | 2 | 1 | 1 | 4
  Serum Glucose Shifts to Low | 1 | 0 | 2 | 3

3. Secondary Outcome: Change in Plasma Concentrations of M-specific A1AT up to 52 Weeks
Description: Change from baseline at Week 52 of plasma concentration of M-specific A1AT for subjects who did not receive PAT post-dose
  Note:
  1. Two subjects in Dose 1 Arm/Group, had results available at Week 52; the remaining 4 subjects in Dose 2 Arm/Group and Dose 3 Arm/Group had resumed PAT therapy after Week 24, and their results were censored from the Week 52 timepoint.
  2. While data on the Total Plasma Concentrations of A1AT up to 52 Weeks were collected for 1 study participant in Part A: Dose 3, no data were collected on the Change in Plasma Concentrations of M-specific A1AT due to the initiation of PAT after 24 weeks in Part A: Dose 3 subjects.
Time Frame: At Week 52
Population: Not analyzed per the statistical analysis plan because participants initiated PAT therapy
Measure: Mean (Standard Deviation); unit: uM
Groups:
- Part A: Dose 1: Single IV infusion at 8E13 total vg
- Part A: Dose 2: Single IV infusion at 4E14 total vg
- Part A: Dose 3: Single IV infusion at 1.2E15 total vg
- Total: All Participants: All subjects who received ADVM-043
Arm/Group | Part A: Dose 1 | Part A: Dose 2 | Part A: Dose 3 | Total: All Participants
Number analyzed (Participants) | 2 | 0 | 0 | 2
uM | 88.050 (19.955) |  |  | 88.050 (19.955)

4. Secondary Outcome: Changes in Total Plasma Concentrations of A1AT up to 52 Weeks
Description: Change from baseline at Week 24 and Week 52 of total A1At plasma concentration for subjects who did not receive PAT post -dose
Time Frame: At Week 52
Population: Not analyzed per the statistical analysis plan because participant initiated PAT therapy
Measure: Mean (Full Range); unit: uM
Groups:
- Part A: Dose 1: Single IV infusion of ADVM-043 8E13 total vg
- Part A: Dose 2: Single IV infusion of ADVM-043 4E14 total vg
- Part A: Dose 3: Single IV infusion of ADVM-043 1.2E15 total vg
- Total: All Participants: All participant who received ADVM-043
Arm/Group | Part A: Dose 1 | Part A: Dose 2 | Part A: Dose 3 | Total: All Participants
Number analyzed (Participants) | 2 | 2 | 2 | 6
uM
  Mean change from Baseline at Week 24 serum Total Protein | 1.230 [-0.08 to 2.54] | 1.870 [0.14 to 3.60] | 1.145 [0.20 to 2.09] | 1.415 [-0.08 to 3.60]
  Mean change from Baseline at Week 52 serum Total Protein: number analyzed (Participants) | 2 | 0 | 1 | 3
  Mean change from Baseline at Week 52 serum Total Protein | 1.220 [-0.44 to 2.88] |  | 0.640 [0.640 to 0.640] | 1.027 [-0.44 to 2.88]

ADVERSE EVENTS:
Time Frame: From ADVM-043 infusion through End-of-Study visit at 52 weeks
Description: Subject incidence of treatment-emergent serious adverse events
Arm/Group | Part A: Dose 1 | Part A: Dose 2 | Part A: Dose 3
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 2/2 | 1/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Dose 1 (N=2) | Part A: Dose 2 (N=2) | Part A: Dose 3 (N=2)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Dose 1 (N=2) | Part A: Dose 2 (N=2) | Part A: Dose 3 (N=2)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Cortisol decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Crystal urine present (Investigations) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrollment was stopped after dosing was complete for participants in Cohorts 1, 2, and 3 of Part A. Cohort 4 of Part A and Part B were not enrolled. Only 6 of the up to 25 potentially anticipated participants were enrolled and received study treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restrictions on the PIs are that Sponsor can review communications by the PI prior to public release and can embargo communications regarding trial results for varying time periods from the time submitted to the sponsor for review. The Sponsor may require changes to the communication after review and may delay publication upon request by the Sponsor to allow the Sponsor to seek/obtain patent protection.

DOCUMENTS (2):
  • Study Protocol (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/86/NCT02168686/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/86/NCT02168686/SAP_001.pdf